CLINICAL TRIAL: NCT01173094
Title: DCLI-II:Optimized Strategy for Diabetic Patients With Critical Limb Ischemia: A Multi-center, Randomized Controlled Trial and Registration Study(Part II)
Brief Title: Optimized Strategy for Diabetic Patients With Critical Limb Ischemia(Part II) (DCLI-II)
Acronym: DCLI-II
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Beijing Tongren Hospital (Other); Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Liu Chang-wei, Vascular Surgery, Peking Union Medical College Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pumch-DCLI-II
Record Dates: First submitted 2010-07-28; First posted 2010-07-30 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2010-07

CONDITIONS: Vascular Diseases; Diabetes
Keywords: Critical limb ischemia; Diabetes Mellitus; Diabetes foot
MeSH Terms: conditions — Vascular Diseases; Diabetes Mellitus; Chronic Limb-Threatening Ischemia | interventions — Angioplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PTA (Experimental): The patients with short-obstruction in the below-knee artery will be included in this group.
  Interventions: Device: Percutaneous Transluminal Angioplasty
- bypass (Experimental): The patients with long-obstruction in the below-knee artery will be included in this group.
  Interventions: Device: below-knee arterial bypass

INTERVENTIONS:
Device: Percutaneous Transluminal Angioplasty — Before operation, take aspirin 100mg every day. During the operation, balloon is delivered by a catheter and positioned through the narrowing in the artery. Then expand the balloon against the wall of the blood vessel to provide a wider channel for blood.
  Arms: PTA
Device: below-knee arterial bypass — Before operation, take aspirin 100mg every day. Perform bypass to below-knee(posterior tibial，anterior tibial or peroneal)arteries, saphenous vein graft with end to side anastomoses
  Arms: bypass

SUMMARY:
The purpose of this trial is to find out the appropriate way to treat DM patients with critical limb ischemia. This trial includes two parts. Part I focuses on the treatment of femoral arterial lesion and part II focuses on the treatment of below-knee arterial lesion.

DETAILED DESCRIPTION:
The trial includes two parts and here is part II. This part is a multi-center, prospective, registration study which focuses on the treatment of below-knee arterial lesion. Totally 130 patients will be entered into this part. They should suffer ischemic symptom with Rutherford 3-6 for the occlusion of the below-knee arteries(anterior tibial、posterior tibial or peroneal artery). According to the lesion length, the patients will accept transluminal angioplasty or below-knee arterial bypass. They will be followed up for 3 years. Study examinations will be done at screening, procedure time, 1, 6, 12, 24 and 36 months after procedure.

ELIGIBILITY:
Inclusion Criteria:

* The patients volunteer to join the trial and sign the formal consent.
* The patients are ≥55 year-old and ≤75 year-old.
* The patients suffer from symptomatic leg ischemia with rutherford classification3, 4 , 5 or 6.
* Obvious stenosis or occlusion in below-knee popliteal artery
* No obvious stenosis or occlusion in the aortoiliac artery; or the lesion could be treated simultaneously or has already been cured.
* No surgical contraindications;no infection in operation region.
* Be diagnosed with DM for at least 1 year.

Exclusion Criteria:

* Refuse random treatment.
* Previous operations on the target artery.
* Acute lower extremity arterial thrombosis.
* Serious major organ failure.
* Allergic to the contrast agent or has contrast nephropathy.
* No clinical compliance or unfit to join the trial

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2010-08; Primary Completion 2013-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Occlusion of the below-knee artery or bypass | 36 months

SECONDARY OUTCOMES:
Mortality | 30 days
  The number of death during the first month after procedure, no matter whether the cause of death is related to the procedure.
Rate of limb salvage | 36 months
Procedural complications, defined as any adverse event | 36 months
  including MI, DVT, hematoma, renal failure, wound infection, lymphatic fistula
Quality of Life assessment | 36 months
  assessment in 1 month,6 months,12 months,24 months and 36 months post procedure
Restenosis measured by Duplex Ultrasound or CTA | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Liu changwei, bachelor, Study Chair
Locations (3):
- China (3):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital, Beijing, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Beijing, Beijing Municipality

REFERENCES:
- See also: the website of the vascular surgery department of PUMCH — http://www.vascular.cn/